CLINICAL TRIAL: NCT01322256
Title: Positron Emission Tomography - Computed Tomography (PET/CT) Scanning for the Follow-up of Antibiotic Treatment of Infectious Osteoarthritis in the Diabetic Foot
Brief Title: PET/CT Scanning for the Follow-up of Antibiotic Treatment of Infectious Osteoarthritis in the Diabetic Foot
Acronym: ISEOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has proven to be infeasible.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AOI/2009/SJ-01; 2010-020160-38 (Other: RCB number)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Foot; Osteoarthritis
MeSH Terms: conditions — Diabetic Foot; Osteoarthritis | interventions — Sulesomab; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Included patients (Experimental): Patients included in the study according to stated inclusion and exclusion criteria
  Intervention: Bone scintigraphy Intervention: Leukoscan Intervention: PET / CT Intervention: Bone biopsy Intervention: Bloodwork
  Interventions: Procedure: Bone scintigraphy; Procedure: Leukoscan; Procedure: PET / CT; Procedure: Bone biopsy; Biological: Bloodwork

INTERVENTIONS:
Procedure: Bone scintigraphy — Bone scintigraphy of the affected area
Procedure: Leukoscan — Scintigraphy with labeled neutrophils
Procedure: PET / CT — PET / CT of the affected area
Procedure: Bone biopsy — A bone biopsy is performed during pre-inclusion work up.
Biological: Bloodwork — CRP and procalcitonin are measured in the pre-inclusion work up.

SUMMARY:
The investigators' primary objective is to assess the predictive power of PET/CT scanning in the evolution of infectious osteoarthritis of the diabetic diabetic after antibiotic therapy prescribed by national and international recommendations.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient has type I or type II diabetes
* Patient consulting in the department of Metabolic and Endocrine Diseases (Caremeau Hospital) or the department of Nutritional Diseases and Diabetology (Grau de Roi Medical Center) at the Nîmes University Hospital
* Patient has infected osteoarthritis of the foot according to the International Working Group on the Diabetic Foot with a probability > 50% (score >= 2).

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* Patient has severe sepsis or a stage 4 infection according to the international consensus on the diabetic foot
* Patient has severe renal insufficiency as defined by glomerular filtration rate < 30ml/min/1.73 m^2, calculated according to the MDRD equation, and is not undergoing dialysis
* Patient has a contra-indication for an MRI
* pacemaker
* intracranial clips
* metallic inclusions
* severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The difference between AUCs for PET/CT scan and scintigraphy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schuldiner, MD, Study Director — Centre Hospitalier Universitaire de Nîmes; Nathalie Jourdan, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - CHU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi